CLINICAL TRIAL: NCT02346695
Title: Vascular and Biochemical Determinants of Left Ventricular Deformation and Twisting-untwisting and Their Interrelation With Aerobic Exercise Capacity in Untreated Arterial Hypertension
Brief Title: Association Between Left Ventricular Deformation and Aerobic Exercise Capacity in Untreated Arterial Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor in Cardiology, University of Athens
Other Study IDs: 214/19-6-12
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Arterial Hypertension
Keywords: LV deformation; Endothelial glycocalyx; Coronary flow reserve
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma in serum for fibrosis and inflammatory markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypertensives: Untreated consecutive patients with newly diagnosed essential hypertension
- Controls: Normotensive individuals

SUMMARY:
Impaired myocardial deformation may determine cardiac diastolic dysfunction. The investigators will investigate the vascular determinants of myocardial deformation and twisting-untwisting and their interrelation with exercise capacity in patients with untreated arterial hypertension

DETAILED DESCRIPTION:
The investigators plan to examine 320 untreated hypertensives and 160 controls. They will measure:

1. the carotid to femoral pulse wave velocity (PWVc) using the Complior apparatus
2. the coronary flow reserve (CFR) at baseline and after adenosine infusion (140 μg x kg-1 x min-1) by Doppler echocardiography
3. the Global Longitudinal strain and strain rate, peak twisting, the percentage changes between peak twisting and untwisting at mitral valve opening (UtwMVO), at peak (UtwPEF) and end of early LV diastolic filling (UtwEDF) by speckle tracking imaging
4. the perfusion boundary region (PBR-micrometers) of the sublingual arterial microvessels (ranged from 5-25 micrometers) using Sideview Darkfield imaging (Microscan, Glycocheck). Increased PBR is considered an accurate non invasive index of reduced endothelial glycocalyx thickness
5. transforming growth factor (TGFb-1), metalloproteinase-9 (MMP-9), markers of collagen synthesis (N-terminal procollagen type-III propeptide , carboxy-terminal propeptide and telopeptide of procollagen type-1, representing cardiac extracellular matrix turnover) and N-terminal pro-brain natriuretic peptide (NT-proBNP) and soluble angiotensin-converting enzyme (sACE).
6. Twenty-four hour daytime and night-time average systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rates as well as 24h-pulse pressure (PP) by means of 24h ambulatory blood pressure monitoring (ABPM) Monitoring will be carried out on the non-dominant arm using the valid recorder TONOPORT V (General Electric, Health Care, Berlin, Germany) after validation of readings against a mercury sphygmomanometer by means of a Y tube. The ABPM device will set to obtain BP readings at 15 min intervals during the day (07.00-23.00) and at 20 min intervals during the night (23.00-07.00). The patients will be instructed to attend their usual day-to-day activities but to keep still at the times of measurements. Recordings will be analysed to obtain
7. oxygen consumption as an absolute value and in relation to body weight (VO2/Kg) and maximum work load (METS) by means of a physician-supervised maximal, symptom-limited cardiopulmonary exercise test (CPET) on a bicycle ergometer using a standard ramping protocol (Oxycon Pro system, Jaeger, Germany).

ELIGIBILITY:
Inclusion Criteria:

* untreated patients with newly diagnosed essential hypertension
* normotensive subjects

Exclusion Criteria:

* history of diabetes
* familiar hyperlipidemia
* coronary CAD
* cardiomyopathy
* chronic pulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 320 ntreated consecutive patients with newly diagnosed essential hypertension and 160 normotensive individuals
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Vascular function in hypertensive and normotensive subjects | Baseline
  Pulse wave velocity by Complior,endothelial glycocalyx thickness by Miscroscan camera and coronary flow reserve by Doppler echocardiography were measured in hypertensive and normotensive subjects
Myocardial deformation in hypertensive and normotensive subjects | Baseline
  Longitundinal, circumferential and radial strain-strain rate were measured by speckle tracking imaging
Left ventricular twisting-untwisting in hypertensive and normotensive subjects | Baseline
  Peak twisting-untwisting ,twisting-untwisting velocity, the percentage difference between peak twisting and untwisting at mitral valve opening , peak and end of early diastolic filling of the left ventricle was measured by speckle tracking imaging

SECONDARY OUTCOMES:
Collagen synthesis in hypertensive and normotensive subjects | Baseline
  Blood levels of N-terminal procollagen type-III propeptide , carboxy-terminal propeptide and telopeptide of procollagen type-1, representing cardiac extracellular matrix turnover were measured in patients with untreated arterial hypertension and normotensive subjects
Inflammation in hypertensive and normotensive subjects | Baseline
  Transforming growth factor b-1, metalloproteinase-9, soluble angiotensin converting enzyme blood levels were measured in patients with untreated arterial hypertension and normotensive subjects
Neurohumoral activation in hypertensive and normotensive subjects | Baseline
  N-terminal pro-brain natriuretic peptide blood levels were measured in patients with untreated arterial hypertension and normotensive subjects
Exercise capacity in hypertensive subjects | Baseline
  Peak oxygen consumption during cardiopulmonary exercise test was measured in patients with untreated arterial hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, Attikon Hospital, University of Athens, Greece; Helen Triantafyllidi, MD, Principal Investigator — 2nd Cardiology Department, Attikon Hospital, University of Athens, Greece; John Lekakis, MD, Principal Investigator — 2nd Cardiology Department, Attikon Hospital, University of Athens, Greece
Locations (1):
- "Attikon" University General Hospital, Haidari, Athens, Attica, Greece

REFERENCES:
- [Derived] Tzortzis S, Ikonomidis I, Triantafyllidi H, Trivilou P, Pavlidis G, Katsanos S, Katogiannis K, Birba D, Thymis J, Makavos G, Varoudi M, Frogoudaki A, Vrettou AR, Vlastos D, Parissis J, Lekakis J. Optimal Blood Pressure Control Improves Left Ventricular Torsional Deformation and Vascular Function in Newly Diagnosed Hypertensives: a 3-Year Follow-up Study. J Cardiovasc Transl Res. 2020 Oct;13(5):814-825. doi: 10.1007/s12265-019-09951-9. Epub 2020 Jan 2. PMID 31898757